CLINICAL TRIAL: NCT05180747
Title: A Randomized Trial of BUrst vs. Spaced Physical Therapy for Parkinson's Disease: The BUS PT Trial
Brief Title: BUrst vs. Spaced Physical Therapy for Parkinson's Disease: The BUS PT Timing Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201903188
Record Dates: First submitted 2021-12-14; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Physical Therapy; Time Up and Go; Spaced Physical Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blinded study. Participants were randomly assigned (1:1) to either burst or spaced groups using a computer random generated sequence. Group allocation could not be hidden from the study participant and thus once baseline measurements were recorded, a disclosure of assignment was made by the study PI. Patients Outcomes measures were be performed at baseline and 6 months by a blinded rater.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Burst group (Other): Patients received two physical therapy sessions weekly for 6 weeks.
  Interventions: Other: Frequency of physical therapy sessions
- Spaced Group (Other): Patients received one physical therapy sessions every 2 weeks for 6 months.
  Interventions: Other: Frequency of physical therapy sessions

INTERVENTIONS:
Other: Frequency of physical therapy sessions — Physical therapy sessions consisted of standard of care practice at our center of excellence i two different frequencies. All patients in both groups received 12 physical therapy sessions. Patients in the burst group received 2 physical therapy sessions per week in 6 weeks, while patients in the spaced group received 1 session every 2 weeks for 6 months.

SUMMARY:
Many patients with Parkinson's Disease (PD) will encounter difficulties with balance, posture, and gait for which physical therapy (PT) has been shown to be beneficial. The purpose of this study is to randomize patients between standard "burst" PT versus "spaced" PT to inform on the optimal frequency of PT for PD patients. Burst PT in this study was defined as 2 PT visits per week for 6 weeks (12 sessions) and spaced PT, as 1 PT visit every other week for 6 months (12 sessions).

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a progressive neurodegenerative disorder with a negative impact on quality of life.1 Many patients with PD will encounter difficulties with balance, posture, transfer, gait and physical capacity due to the motor symptoms of the disease.2 For these symptoms, physical therapy (PT) has been shown to be beneficial and clinically useful for the motor symptoms and thus is routinely prescribed alongside medical management. However, despite increasing evidence of the positive effects of physical therapy for patients with PD, there is no standard approach for organizing physiotherapy in the context of multidisciplinary care. Administration of physical therapy as a "burst" of frequent sessions delivered over 4-6 weeks is the most commonly employed strategy in PD patients and is driven largely by the payer system. Burst therapy has been useful in post-stroke and post traumatic brain injury rehabilitation, however, the investigators of this study hypothesize that this approach will be suboptimal in PD when compared to therapy which is "spaced" over a longer period of time. The purpose of this study is to randomize patients between typical "burst" PT versus "spaced" PT to inform on the optimal frequency of PT for PD patients. Burst PT in this study was defined as 2 PT visits per week for 6 weeks (12 sessions) and spaced PT, as 1 PT visit every other week for 6 months (12 sessions).

30 PD patients were recruited as part of a pilot trial to assess the effectiveness of burst vs. spaced physical therapy (the BUS PT trial). Baseline measures were collected on all patients, including the timed up and go test (TUG), the baseline frequency of utilization of PT, falls, fractures, hospitalizations, the 10 meter walk test (10MWT), the Mini Balance Evaluation Systems Test (miniBESTest), objective gait analysis using Gaitrite, the Parkinson's Disease Questionnaire-39 (PDQ39), the Unified Parkinson's Disease Rating Scale (UPDRS) "ON" and "OFF" motor scores, the quantitation of the levodopa equivalent daily doses (LEDD), and the Godin Leisure Activity Questionnaire to assess baseline exercise levels.

The investigators hypothesized that "spaced" PT is beneficial for maintenance of physical function in PD. Prior collective evidence suggests that long-term continuous exercise in PD patients is associated with positive outcomes, however a spaced PT approach has not been employed. This study will provide useful data that will directly impact payer systems, reimbursements and access to care for PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-90 years
* Parkinson's disease as measured by Hoehn & Yahr stage 2-3
* Idiopathic Parkinson's Disease patients diagnosed by a Movement Disorder Neurologist
* Stable dopaminergic medication for 1 month prior to the study and during the study (6 month intervention)
* Requires ongoing physical therapy as assessed by a physical therapist

Exclusion Criteria:

* Comorbidities including orthopedic injuries or cardiopulmonary disease that would potentially interfere with physical therapy and assessments
* Severe cognitive impairments (MMSE <21)
* Unable to participate in all therapy sessions

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change between baseline and 6-month Timed Up and Go test (TUG) | Baseline up to 6-month follow up
  The TUG test is a validated and reliable tool to assess balance and mobility in Parkinson's disease. It has been used as an outcome measure in many trials involving PT and exercise in PD and is frequently included in standard PT visits. Patients wear their regular footwear and can use a walking aid, if needed. Patient starts the test sitting back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor. Once examiner says go. the patient has to get up from the chair, walk until the line on the floor, come back and sit down on the chair. Timing begins when examiner says "go" and stops after patients sits back down. An older adult that takes 12 or more seconds to complete the task is at risk for falling.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) motor score | Baseline up to 6-month follow up
  Minimum value for UPDRS part III is 0 and maximum value is 27. High scores mean a worse outcome.
The Mini Balance Evaluation Systems Test (MiniBesTest) | Baseline up to 6-month follow up
  The MiniBesTest assesses dynamic balance: anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. It is a 14-item test scored on a 3 level ordinal scale. Minimum score is 0 and maximum score is 32. High scores mean better outcome.
10 meter walk test (10MWT) | Baseline up to 6-month follow up
  This a performance measure used to assess walking speed in meters per second over a short distant.
Non-motor symptoms PD questionnaire (NMS) | Baseline up to 6-month follow up
  NMS is a screening questionnaire comprising 30 items. It was not designed as a quantitative scale, however, a total score for the questionnaire is calculated by summing all the positive ("yes") responses. Minimum score is 0 and maximum score is 30. High scores correlate to worse outcomes. PD patients have higher scores when compared to control patients.
Parkinson's Disease Questionnaire-39 (PDQ39) | Baseline up to 6-month follow up
  PDQ39 is a 39-item self reported questionnaire that assesses PD-specific health related quality over the last month. It assesses the 8 quality of life dimensions: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication and bodily discomfort. Minimum score is 0 and maximum score is 156. High scores mean worse outcomes.
Levodopa equivalent daily doses (LEDD) | Baseline up to 6-month follow up
  Conversion factor to generate a total Levodopa equivalent daily dose (LEDD), calculated as a sum of each parkinsonian medication. LEDD provides an artificial summary of the total daily medication a patient is receiving .
Baseline frequency of utilization of PT | Baseline up to 6-month follow up
  Frequency of PT sessions patients were having before starting the study.
Objective gait analysis using Gaitrite | Baseline up to 6-month follow up
  Patients walk on a 3m walking mat embedded with 256 sensors that are triggered when pressure is applied. The GAITRite system automates measuring temporal (timing) and spatial (distance) gait parameters (temporal/spatial) and 8 levels of relative pressure. Data are processed by a second compatible computer by using GaitMat software.
Falls diary | Baseline up to 6-month follow up
  It consists in one way of recording fall frequency and the surrounding circumstances. Patients are encouraged to recall and identify the key circumstances surrounding falls.
Godin Leisure Activity Questionnaire | Baseline up to 6-month follow up
  Patients have to disclose how many times on the average typical 7-Day period (a week) they do the following kinds of exercise for 15 or more minutes: STRENUOUS EXERCISE (HEART BEATS RAPIDLY) (e.g., running, jogging, hockey, football, soccer, squash, basketball, cross country skiing, judo, roller skating, vigorous swimming, vigorous long distance bicycling); MODERATE EXERCISE (NOT EXHAUSTING) (e.g., fast walking, baseball, tennis, easy bicycling, volleyball, badminton, easy swimming, alpine skiing, popular and folk dancing) and MILD/LIGHT EXERCISE (MINIMAL EFFORT) (e.g., yoga, archery, fishing from river bank, bowling, horseshoes, golf, snow-mobiling, easy walking). Weekly leisure activity score = (9 × Strenuous) + (5 × Moderate) + (3 × Light). Minimum score is 0. Maximum score is 119. High scores mean that the patient is more active. Patients can be classified as sedentary (<14), moderately active (14-23) and active (24 or more).
Change between 6-week and 6-month Timed Up and Go test (TUG) | 6-week follow up (burst group only) and 6-month follow up
  The TUG test is a validated and reliable tool to assess balance and mobility in Parkinson's disease. It has been used as an outcome measure in many trials involving PT and exercise in PD and is frequently included in standard PT visits. Patients wear their regular footwear and can use a walking aid, if needed. Patient starts the test sitting back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor. Once examiner says go. the patient has to get up from the chair, walk until the line on the floor, come back and sit down on the chair. Timing begins when examiner says "go" and stops after patients sits back down. An older adult that takes 12 or more seconds to complete the task is at risk for falling.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Loong Kelvin Au, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices), study protocol and statistical analysis plan will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be submitted up to 36 months following article publication. After 36 months, data will be available in our University's data warehouse, but without investigator support other than deposited metadata. Proposals should be directed to janinelobolopes@ufl.edu.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal